CLINICAL TRIAL: NCT04348526
Title: The Effect of Corticision on Perceived Pain and Discomfort for Patients With Crowded Lower Anterior Teeth: Randomized Clinical Trial
Brief Title: Evaluation of the Levels of Pain and Discomfort Between Two Methods of Leveling and Alignment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-03-2020
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Crowding
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticision (Experimental): Patients will undergo a corticision procedure in order to accelerate tooth movement
  Interventions: Procedure: Corticision
- Traditional treatment (Active Comparator): Patients will undergo traditional orthodontic treatment without any surgical intervention.
  Interventions: Procedure: Traditional orthodontic treatment

INTERVENTIONS:
Procedure: Corticision — Surgical intervention is going to be used in the interdental areas between the lower anterior teeth to accelerate tooth movement. Three incisions are going to be made
  Arms: Corticision
Procedure: Traditional orthodontic treatment — No surgical intervention will be used, just normal orthodontic sequence of procedures.
  Arms: Traditional treatment

SUMMARY:
The duration of orthodontic treatment is one of the exacerbation causes of orthodontic pain. Several methods have been suggested to reduce the duration of orthodontic treatment classified to surgical and non-surgical methods.

Researches used minimally invasive surgical methods like corticision, piezocesion, micro-osteoperforation, and piezo-puncture indicated that most of these methods can accelerate dental movement by 20 - 40% without causing additional pain as a result of using those methods. Applying corticision on the lower anterior teeth using a surgical blade and a hammer may accelerate tooth alignment during orthodontic treatment. This study consists of two groups, patients will be randomly assigned to one of these two groups.

DETAILED DESCRIPTION:
Pain is defined as an unpleasant emotional sensory experience associated with actual or potential harm. It was mentioned as one of the most common complaints related to orthodontic treatment, and around 65-95% of patients undergoing orthodontic treatment suffer from various degrees of pain.

Corticision is one of the minimally invasive surgical procedures that is not associated with flap lifting. It was used to accelerate tooth movement in animals and case report studies. Its application on humans may aggravate their fear and anxiety towards the pain that may accompany this technique.

No study in the literature has been searched in patient perception of pain, discomfort, levels of acceptance and satisfaction accompanied corticision application, but in this study, these previous variables accompanied corticision technique have been studied on crowded lower anterior teeth cases which are one of the most common types of malocclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 24 years
2. Completion permanent dentition (except third molars)
3. Mild to moderate crowding (2-6 mm according to Little's index)
4. Absence of medications intake that interferes with pain perception for at least one week before the beginning of the treatment

Exclusion Criteria:

1. Systematic diseases that could affect bone and tooth movement and no contraindication avoid oral surgery
2. Medical conditions that affect tooth movement (Corticosteroid, NSAIDs)
3. Patients had previous orthodontic treatments
4. Poor oral hygiene or concurrent periodontal disease

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change in the Perception of Pain | At 24 hours following the onset of treatment (bonding of the appliance), then at 7 days, 14 days following the onset of orthodontic treatment
  Pain is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of pain being experienced. The left end of the line refers to no pain (VAS=0) where the right end refers to maximum (unimaginable) pain (VAS=100). The level of pain is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the pain.
Change in the Perception of Discomfort | At 24 hours following the onset of treatment (bonding of the appliance), then at 7 days, 14 days following the onset of orthodontic treatment
  Discomfort is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of discomfort being experienced. The left end of the line refers to no discomfort (VAS=0) where the right end refers to maximum discomfort (VAS=100). The level of discomfort is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the discomfort.
Change in the Perception of Swelling | At 24 hours following the onset of treatment (bonding of the appliance), then at 7 days, 14 days following the onset of orthodontic treatment
  Swelling is assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of swelling being experienced. The left end of the line refers to no swelling (VAS=0) where the right end refers to maximum swelling (VAS=100). The level of swelling is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the swelling
Change in the Levels of Difficulties in Mastication | At 24 hours following the onset of treatment (bonding of the appliance), then at 7 days, 14 days following the onset of orthodontic treatment
  Difficulties of mastication are assessed by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of difficulties in mastication being experienced. The left end of the line refers to no difficulties (VAS=0) where the right end refers to maximum difficulties (VAS=100). The level of difficulties in mastication is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the difficulties of mastication.
Analgesic Consumption | The 7th day following the onset of treatment (i.e. at the second visit of the patients following his orthodontic appliance bonding; one-time assessment)
  Patients in both groups were asked about taking analgesics and their quantity (mg) They answered about taking analgesics using a two-point scale (1. Yes or 2. No), and their quantity by mentioning how many tablets they took.

SECONDARY OUTCOMES:
Patients' satisfaction | At the end of leveling and alignment which is expected to occur within 4 to 6 months
  Satisfaction is assessed for both groups by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of satisfaction. The left end of the line refers to no satisfaction (VAS=0) where the right end refers to maximum satisfaction (VAS=100). The level of satisfaction is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the satisfaction.
Ease of the procedure | At the end of leveling and alignment which is expected to occur within 4 to 6 months
  Procedure's easiness is assessed for both groups by asking the study participant to place a mark on a horizontal 100 mm line to indicate the level of ease. The left end of the line refers to no ease (VAS=0) where the right end refers to maximum ease (VAS=100). The grade of ease is represented in the number of millimeters measured from the left end of the line to the mark pointed out by the patient. This is called the Visual Analogue Score (VAS) where the higher the number is the more intense the ease of the procedure.
The possibility of repeating the procedure | At the end of leveling and alignment which is expected to occur within 4 to 6 months
  Patients in the corticision group will be asked about the possibility of repeating the procedure if they had the chance to give their decision again. The answer will be collected using a two-point scale (1. Yes or 2. No).
Recommendation to a friend | At the end of leveling and alignment which is expected to occur within 4 to 6 months
  Patients in the corticision group will be asked about if they would recommend this procedure to a friend. The answer will be collected using a two-point scale (1. Yes or 2. No).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Radwan Sirri, DDS MSc, Principal Investigator — MSc student in Orthodontics, University of Damascus Dental School; Ahmad S Burhan, DDS MSc PhD, Study Chair — Professor of Orthodontics, University of Damascus, Damascus, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Professor of Orthodontics, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- Orthodontic Department, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984
- [Background] Alkebsi A, Al-Maaitah E, Al-Shorman H, Abu Alhaija E. Three-dimensional assessment of the effect of micro-osteoperforations on the rate of tooth movement during canine retraction in adults with Class II malocclusion: A randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2018 Jun;153(6):771-785. doi: 10.1016/j.ajodo.2017.11.026. PMID 29853235
- [Background] Charavet C, Lecloux G, Bruwier A, Rompen E, Maes N, Limme M, Lambert F. Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res. 2016 Aug;95(9):1003-9. doi: 10.1177/0022034516645066. Epub 2016 Apr 29. PMID 27129491
- [Background] Uribe F, Davoody L, Mehr R, Jayaratne YSN, Almas K, Sobue T, Allareddy V, Nanda R. Efficiency of piezotome-corticision assisted orthodontics in alleviating mandibular anterior crowding-a randomized clinical trial. Eur J Orthod. 2017 Nov 30;39(6):595-600. doi: 10.1093/ejo/cjw091. PMID 28371882
- [Background] Yavuz MC, Sunar O, Buyuk SK, Kantarci A. Comparison of piezocision and discision methods in orthodontic treatment. Prog Orthod. 2018 Oct 29;19(1):44. doi: 10.1186/s40510-018-0244-y. PMID 30370430